CLINICAL TRIAL: NCT01965990
Title: A 2-week Course of Enteral Treatment With a Very Low-calorie Protein-based Formula for the Management of Severe Obesity
Brief Title: VLCD by Enteral Route for Weight Loss
Acronym: NEP
Status: Completed | Type: Observational
Sponsor: San Giuseppe Moscati Hospital (Other)
Responsible Party: Principal Investigator, Giuseppe Castaldo, Medical Doctor, Director of the Clinical Nutrition Unit, San Giuseppe Moscati Hospital
Other Study IDs: 23bis
Record Dates: First submitted 2013-10-16; First posted 2013-10-18 (Estimated); Last update posted 2013-10-22 (Estimated); Status verified 2013-10

CONDITIONS: Severe Obesity
Keywords: Enteral nutrition; very low-calorie diet; severe obesity; weight loss; ketosis
MeSH Terms: conditions — Obesity, Morbid; Weight Loss; Ketosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- NEP: Patients undergoing the administration of a homemade very low-calorie protein-based formula (2000 mL per day) by enteral route for 14 days
  Interventions: Other: NEP

INTERVENTIONS:
Other: NEP — A homemade very low-calorie protein-based formula by enteral route (8-French nasogastric tube) for 14 days. The administration was continuous (h-24) by a feeding pump. The formula was made up of a fixed amount of aminoacids and a variable amount of high-quality proteins: 1.2 g/kg (ideal body weight). Other components were: pro-lipolytic substances (coenzyme Q10 and L-carnitine), linseed oil, policosanol, fructo-oligo saccharides, potassium, sodium and magnesium chloride. The intervention included also the daily oral administration of a multivitamin-multimineral supplement, alkalizing substances (calcium carbonate, 1500 mg; magnesium carbonate, 850 mg; potassium bicarbonate, 500 mg; sodium bicarbonate, 1500 mg; potassium citrate, 500 mg) and herbal remedies. All patients were also prescribed treatment with a proton pump inhibitor and ursodeoxycholic acid. A minimum intake of 2 liters/day of unsweetened fluids was recommended (3 litres in case of a history of kidney stones).

SUMMARY:
Body weight excess, from overweight to overt obesity, is associated with adverse health outcomes. In view of the time-trends of the obesity epidemic and the related cost burden, the search for effective strategies for weight reduction and long-term maintenance of weight loss (WL) is at the top of the agenda of public health systems.

The current first-line strategy includes several treatment options and dietary interventions to be implemented together with an exercise program. Unfortunately, compliance with intervention in the long-term is difficult. It is not infrequent to observe people following one diet after another and experiencing multiple failures which, in turn, lead to higher body weight and adverse consequences on body composition and fat distribution. The higher the number of attempts, the more difficult the adherence to further interventions. In the presence of severe (body mass index >40 kg/m2) or complicated obesity, bariatric surgery could be proposed. This therapeutic option is effective, but is not devoid of complications and may be irreversible. Obesity-related complications, such as diabetes, hypertension or sleep apnoea are likely to occur more frequently with increasing body mass index (BMI) and rapid and considerable WL is mandatory to curtail such risks.

In this scenario, alternative treatment options are warranted. About 40 years ago, after the introduction of protein-sparing modified fasting (PSMF) achieved through the use of oral high-protein foods or liquid formula diets by Blackburn and Bistrian, several studies evaluated its effectiveness and safety. They showed that responsible and supervised very-low calorie diets (VLCDs) could be considered safe and appropriate therapy for obesity.

The purpose of the present study was to investigate the potential role of a 2-week course of enteral treatment with a very low-calorie protein-based formula in the management of severe obesity.

The rationale of this treatment option rests on the following considerations: 1) VLCDs appear to be able to reduce cardiovascular risk rapidly and effectively; 2) VLCDs induce considerable short and long-term WL; 3) optimal compliance with the intervention, as active participation of the patient is not required; 4) continuous administration of the intervention formula by enteral route enables the the maintenance of the body amino acid pool.

Before being proposed for clinical use, a new WL program should be scientifically evaluated. Accordingly, in the present study, attention was focused not only on efficacy in terms of improving the cardiometabolic risk profile, but also on the feasibility and safety of the procedure.

ELIGIBILITY:
Inclusion Criteria:

* age >=18 years
* severe obesity (body mass index [BMI] >=40 kg/m2)
* history of multiple failures in weight loss programs

Exclusion Criteria:

* age >=70 years
* insulin-dependent diabetes mellitus
* a psychiatric disorder
* previous (<1 year since last chemo- or radiotherapy) neoplastic disease
* current neoplastic disease
* established vascular disease
* recent (6 months), history of diet-induced or unintentional weight loss
* moderate-to-severe heart failure
* arrhythmia
* renal failure (creatinine >1.5 mg/dL)
* current hepatitis
* liver cirrhosis
* any type of gastrointestinal disease
* moderate-severe hypoalbuminemia (<3.0 g/dL)
* altered serum electrolytes
* any other contra-indication to enteral nutrition
* refusal to give written informed consent

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive severly obese patients attending the Clinical Nutrition Unit of our institution for a weight loss program
Sampling Method: Non-Probability Sample
Enrollment: 364 (Actual)
Dates: Start 2010-04; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Weight loss | 14 days
  Percentage of weight loss
Feasibility | 14 days
  Necessity to discontinue the intervention
Safety | 14 days
  Frequency of the following side effects: asthenia, headache, dizziness, fainting, orthostatic hypotension, heartburn, nausea, vomiting, palpitations, muscle cramps, hunger, constipation. evaluation of changes in the following hematological and biochemical parameters and, for those presenting with normal values, by the excursion outside of the reference ranges of our laboratory (new cases): hemoglobin, total lymphocyte count, urea, creatinine, uric acid, albumin, serum enzymes (cholinesterase, transaminases, γ-glutamyl-transferase, serum creatine phosphokinase and serum lactate dehydrogenase ) and electrolytes (sodium, potassium, magnesium, calcium and phosphorus).

SECONDARY OUTCOMES:
Anthropometric and biochemical parameters | 14 days
  Changes (increase [high density cholesterol, apolipoprotein A-I and growth hormone] or more frequently reduction [all the others]) in the following study parameters: body mass index, waist circumference, hip circumference, waist-hip ratio, uric acid, glucose, insulin, insulin resistance, C-peptide, glycosylated hemoglobin, insulin-like growth factor 1, total cholesterol, high density cholesterol, low density cholesterol, triglycerides, triglyceride/high density cholesterol ratio, apolipoprotein B, apolipoprotein B/apolipoprotein A-I ratio, transaminases, γ-glutamyl-transferase.

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe Castaldo, MD, Principal Investigator — Clinical Nutrition Unit - A.O.R.N. "San Giuseppe Moscati", Avellino, Italy
Locations (1):
- Clinical Nutrition Unit - A.O.R.N. "San Giuseppe Moscati", Avellino, Avellino, Italy

REFERENCES:
- [Derived] Castaldo G, Monaco L, Castaldo L, Sorrentino P. A 2-Week Course of Enteral Treatment with a Very Low-Calorie Protein-Based Formula for the Management of Severe Obesity. Int J Endocrinol. 2015;2015:723735. doi: 10.1155/2015/723735. Epub 2015 May 6. PMID 26064113